CLINICAL TRIAL: NCT04481139
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Adaptive Seamless Phase 2/3 Clinical Study to Evaluate the Efficacy and Safety of SHR0302 in Active Ankylosing Spondylitis Subjects
Brief Title: A Study to Evaluate the Efficacy and Safety of SHR0302 in Patients With Ankylosing Spondylitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHR0302-302
Record Dates: First submitted 2020-07-15; First posted 2020-07-22 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2022-07

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — ivarmacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SHR0302 dose1 (Experimental): SHR0302 dose1 for 24 weeks
  Interventions: Drug: SHR0302
- SHR0302 dose2 (Experimental): SHR0302 dose2 for 24 weeks
  Interventions: Drug: SHR0302
- SHR0302 dose3 (Experimental): SHR0302 dose3 for 24 weeks
  Interventions: Drug: SHR0302
- Placebo (Placebo Comparator): Placebo for 12 weeks
  Interventions: Drug: SHR0302 placebo

INTERVENTIONS:
Drug: SHR0302 — SHR0302, oral, once daily
  Arms: SHR0302 dose1; SHR0302 dose2; SHR0302 dose3
Drug: SHR0302 placebo — SHR0302 placebo, oral, once daily
  Arms: Placebo

SUMMARY:
This study is to evaluate the efficacy and safety of different doses of JAK1 inhibitor SHR0302 in subjects with active ankylosing spondylitis.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed informed consent.
* AS diagnosis consistent with the Modified New York Criteria for AS (1984);
* Participant must have baseline disease activity as defined by having a Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score >= 4 and a Patient's Assessment of Total Back Pain score >= 4 based on a 0 - 10 Numeric Rating Scale (NRS) at the Screening and Baseline Visits.
* Participant has had an inadequate response to at least two Nonsteroidal Anti-inflammatory Drugs (NSAIDs) over an at least 4-week period in total at maximum recommended or tolerated doses, or participant has an intolerance to or contraindication for NSAIDs as defined by the Investigator.
* If subjects are taking permitted csDMARDs or low-dose corticosteroid orally at baseline , the stable doses should have lasted for more than 4 weeks already.
* BMI ≥18 kg/m2

Exclusion Criteria:

* Pregnant women or refuse to receive contraception during the study.
* Lab abnormality within 4 weeks of randomization as follows: WBC count <3.0×10^9/L；neutrophil count<1.5×10^9/L;hemoglobin level<90.0 g/L ; platelet count <100×10^9/L; AST or ALT levels greater than the upper limit of normal; HBsAg or HCV or HIV antibody positivity.
* History of other autoimmune diseases ; history of cancer or infection including tuberculosis and hepatitis; history of important cardiovascular events or thrombotic diseases.
* Previous treatment with JAK inhibitor or cytotoxic drugs; bDMARDs within 6 months of randomization; other strong immunosuppressants within 6 months of randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Assessment in Ankylosing Spondylitis (ASAS) 20 response at Week 12. | Week 12
  ASAS20 is defined as a >= 20% improvement and an absolute improvement of >= 1 units (on a scale of 0 to 10) from Baseline in at least 3 of the 4 domains (patient's global assessment, back pain, function and inflammation) with no deterioration in the remaining domain (where deterioration is defined as a worsening of >= 20% and a net worsening of >= 1 unit [on a scale of 0 to 10])

SECONDARY OUTCOMES:
Percentage of Participants with Assessment in Ankylosing Spondylitis (ASAS) 20 response at Week 24. | Week 24
  ASAS20 is defined as a >= 20% improvement and an absolute improvement of >= 1 units (on a scale of 0 to 10) from Baseline in at least 3 of the 4 domains (patient's global assessment, back pain, function and inflammation) with no deterioration in the remaining domain (where deterioration is defined as a worsening of >= 20% and a net worsening of >= 1 unit [on a scale of 0 to 10]) at Week 24.
Percentage of Participants with Assessment in Ankylosing Spondylitis (ASAS) 40 response at Week 12 and Week 24. | Week 12 and Week 24
  ASAS40 is defined as a >= 40% improvement and an absolute improvement of ≥ 2 units (on a scale of 0 to 10) from Baseline in at least 3 of the 4 domains (patient's global assessment, back pain, function and inflammation) with no worsening at all in the remaining domain.
Percentage of Participants with Assessment in Ankylosing Spondylitis (ASAS) 5/6 response at Week 12 and Week 24. | Week 12 and Week 24
  ASAS5/6 is defined as an improvement of at least 20 % in at least five of these six domains (patient global, pain, function, inflammation, CRP, and spinal mobility).
Change from baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Week 12 and Week 24
  BASDAI is a commonly used measure to define disease activity levels in axSpA patients. It consists of 6 questions on a 0 through 10 numeric rating scale (NRS) (0 being no problem and 10 being the worst problem) pertaining to the 5 major symptoms of AS: Fatigue, Spinal pain, Joint pain/swelling, Areas of localized tenderness, Morning stiffness duration, and Morning stiffness severity.
Change from baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) at Week 12 and Week 24. | Week 12 and Week 24
  The BASFI is a validated patient reported outcome (PRO) instrument for use in the AS patient population. It consists of 10 items measured on a 0 to 10 NRS, which assesses the ability to perform activities known to be problematic to AS patients such as dressing, bending, reaching, turning, and climbing steps. The total scores range from 0 to 10.
Change from baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI) at Week 12 and Week 24. | Week 12 and Week 24
  The BASMI will be conducted at the visits specified to evaluate spinal mobility in a participan.
Change from baseline in Short-Form-36-Health Survey (SF-36) at Week 12 and Week 24. | Week 12 and Week 24
  SF-36 is a standardized survey evaluating 8 aspects of functional health and wellbeing: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (0=no functioning, 100=highest level of functioning). Missing data at Week 12 were imputed by LOCF if data at an early visit (discontinuation visit) were available.
Change from baseline in Ankylosing Spondylitis Quality of Life (ASQoL) at Week 12 and Week 24. | Week 12 and Week 24
  The ASQoL is an 18-item axSpA-specific Quality of Life (QoL) PRO measure validated in the AS patient population. Concepts measured include activities of daily life, emotional functioning, pain, fatigue, and sleep problems. Each item on ASQoL is given a score of "1" or "0," where a score of "1" is given when an item is affirmed indicating adverse QoL. Total scores can range from 0 (good QoL) to 18 (poor QoL).

CONTACTS AND LOCATIONS:
Locations (1):
- Zhanguo Li, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Xu X, Wei H, Liu L, Yang R, Shi Q, Pang D. Ivarmacitinib improves patient-reported outcomes across multiple domains in patients with active ankylosing spondylitis: a post hoc analysis of a phase II/III trial. Front Pharmacol. 2025 Nov 20;16:1710434. doi: 10.3389/fphar.2025.1710434. eCollection 2025. PMID 41357869